CLINICAL TRIAL: NCT05447234
Title: Exploratory Clinical Study of TCRx_T Cells in the Treatment of Advanced or Recurrent Gastric/Gastroesophageal Junction Cancer After Failure of First Chemotherapy
Brief Title: TCRx_T Cells for Advanced or Recurrent Gastric/Gastroesophageal Junction Cancer After Failure of First Chemotherapy
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: TCRx Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSH02-TCRXT-CJ
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer
Keywords: T Cell Receptor; Gastric Cancer; Gastroesophageal-junction Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: ① 1x10^7/m2
  * 3x10^7/m2；
    * 1x10^8/m2；
      * 3x10^8/m2；
        * 1x10^9/m2。
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCRX-T (Experimental): ① 1x10^7/m2 ;
  * 3x10^7/m2；
    * 1x10^8/m2；
      * 3x10^8/m2；
        * 1x10^9/m2。
  Interventions: Biological: Tcrx T cell

INTERVENTIONS:
Biological: Tcrx T cell — Sequential IV infusion

SUMMARY:
To observe and determine the safety, tolerability, cellular pharmacokinetics and efficacy of TCRx T cells in patients with advanced or recurrent gastric/gastroesophageal junction cancer after failure of first chemotherapy.

DETAILED DESCRIPTION:
1. Sign the informed consent for clinical trials
2. Subject screening
3. Extract the blood of the subjects and isolate the PBMC
4. Find a patient-specific tumor-specific TCR sequence combination, which is a multi-targeted tumor-specific combination.
5. Transfer of personalized tumor-specific TCRs into patient autologous CD8 T cells by gene editing
6. Large-scale culture and expansion of gene-edited T cells
7. T cell viability, infection efficiency and microbial detection in hospital
8. Calculate the number of cells in the patient's body according to TCRx T
9. Injecting TCRx T cells back into the subject
10. Within 7 days after the injection, the subject's post-dose reaction should be closely observed in the hospital
11. After the first injection, continue to reinfuse TCRx T cells up to 4 times according to the treatment effect and the incidence of adverse events, and be hospitalized after each injection to closely monitor possible adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old;
2. Histologically confirmed advanced/locally advanced or metastatic gastric cancer at the stomach or gastroesophageal junction, progressed after first-line chemotherapy, or recurrence after gastric/gastroesophageal junction surgery combined with neoadjuvant/adjuvant chemotherapy
3. Expected survival time ≥ 3 months
4. Eastern Cooperative Oncology Group (ECOG) score 0-2
5. According to the Response Evaluation Criteria for Solid Tumors (RECIST 1.1), at least one one-dimensional, measurable tumor (short-axis diameter greater than 1 cm)
6. Normal bone marrow hematopoietic function: (leukocytes≥4000 cells/㎕, neutrophils≥1500 cells/㎕, platelet counts≥100000 cells/㎕)
7. Normal liver and kidney function: serum bilirubin <1.5mg/dl, AST (SGOT) and ALT (SGPT) <2.5UNL, alkaline phosphatase <5UNL; serum creatinine <1.5mg/dl;
8. Men and women must take appropriate contraceptive measures.

Exclusion Criteria:

1. Patients with previous non-gastric/gastroesophageal junction malignant tumor
2. History of severe acute allergy
3. There is an uncontrolled infection
4. History or clinical evidence of central nervous system (CNS) metastasis or leptomeningeal carcinomatosis
5. History of cerebrovascular accident within the past 6 months, including transient ischemic attack (TIA), pulmonary embolism or untreated deep vein thrombosis (DVT)
6. History of one or more of the following cardiovascular diseases within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass grafting, symptomatic peripheral vascular disease , NYHA type III or IV congestive heart failure
7. Poor control of hypertension
8. QT interval >480ms
9. Evidence of active bleeding or bleeding tendency
10. Clinically significant gastrointestinal abnormalities, such as bleeding, obstruction, and high risk of perforation
11. Grade 3 or 4 diarrhea
12. Any serious and/or unstable previous medical, psychiatric, or other circumstances that may affect subject safety, provide informed consent, or comply with research procedures
13. Unable or unwilling to stop using illicit drugs for at least 14 days or drug half-life (whichever is longer) before and during the first study drug administration
14. Treated with any of the following anticancer therapies: radiotherapy, tumor embolization or chemotherapy, immunotherapy, biological therapy within 14 days before the first dose; neoadjuvant chemotherapy or adjuvant chemotherapy must be at least 6 months before the start of the study Finish
15. Any persistent toxicity greater than grade 1 and/or worsening in severity from prior anticancer therapy, except for alopecia
16. Participate in a clinical trial of another investigational drug within 30 days prior to the start of the study
17. Pregnant or lactating women
18. Men or women planning to become pregnant within the next six months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
tumor volume | about 2 years
  RECIST 1.1
Overall Survival | about 2 years
  The time from randomization to death due to any reason.

SECONDARY OUTCOMES:
AEs | about 2 years
  CTCAE5.0